CLINICAL TRIAL: NCT00433966
Title: Dual Arm Factorial Randomized Trial in Patients w/ST Segment Elevation AMI to Compare the Results of Using Anticoagulation With Either Unfractionated Heparin + Routine GP IIb/IIIa Inhibition or Bivalirudin + Bail-out GP IIb/IIIa Inhibition; and Primary Angioplasty With Stent Implantation With Either a Slow Rate-release Paclitaxel-eluting Stent (TAXUS™) or Uncoated Bare Metal Stent (EXPRESS2™)
Brief Title: Harmonizing Outcomes With Revascularization and Stents in Acute Myocardial Infarction
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cardiovascular Research Foundation, New York (Other)
Collaborators: Boston Scientific Corporation (Industry); The Medicines Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: HORIZONS AMI
Record Dates: First submitted 2007-02-09; First posted 2007-02-12 (Estimated); Results first posted 2017-12-04 (Actual); Last update posted 2017-12-04 (Actual); Status verified 2017-11

CONDITIONS: Myocardial Infarction
Keywords: Myocardial Infarction; Angioplasty; Myocardial Ischemia; Myocardial Reperfusion; Stents; Heart Disease
MeSH Terms: conditions — Myocardial Infarction; Myocardial Ischemia; Heart Diseases | interventions — bivalirudin; Heparin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pharmacology Arm (Active Comparator): To establish the safety and efficacy of the use of bivalirudin in patients with acute myocardial infarction undergoing a primary angioplasty strategy by showing that compared to unfractionated heparin plus routine use of GP IIb/IIIa inhibitors, bivalirudin (with use of GP IIb/IIIa inhibitors reserved for angioplasty complications) results in:
  1. reduced rates of major bleeding events at 30 days
  2. similar rates of major adverse ischemic cardiac events at 30 days
  3. reduced rates of the composite of major adverse ischemic cardiac events + major bleeding at 30 days.
  Interventions: Drug: Bivalirudin; Drug: Unfractionated heparin
- Stent Arm (Active Comparator): To establish the safety and efficacy of the paclitaxel-eluting TAXUS™ stent by showing that compared to an otherwise identical bare metal EXPRESS2™ stent, the TAXUS™ stent results in:
  1. reduced rates of target lesion revascularization for ischemia at 1 year
  2. similar rates of death, reinfarction, stroke or stent thrombosis at 1 year
  3. lower rates of analysis segment binary angiographic restenosis at 13 months
  Interventions: Device: Bare metal stent; Device: Paclitaxel-eluting stent

INTERVENTIONS:
Drug: Bivalirudin — Bivalirudin bolus of 0.75 mg/kg IV, followed by an infusion of 1.75 mg/kg/h as soon as logistically feasible (ideally in the emergency room).
  Other Names: Angiomax
  Arms: Pharmacology Arm
Drug: Unfractionated heparin — 60 U/kg of IV heparin, started as soon as possible (ideally in the emergency room).
  Other Names: Heparin Sodium
  Arms: Pharmacology Arm
Device: Bare metal stent — Uncoated bare metal stent
  Other Names: EXPRESS2™
  Arms: Stent Arm
Device: Paclitaxel-eluting stent — slow rate-release paclitaxel-eluting stent
  Other Names: TAXUS™
  Arms: Stent Arm

SUMMARY:
The primary objectives of the trial are:

1. To establish the safety and efficacy of the use of bivalirudin (+ bail-out GP IIb/IIIa inhibitors) compared to the use of unfractionated heparin + GP IIb/IIIa inhibitors in patients with acute myocardial infarction undergoing a primary angioplasty strategy.
2. To establish the safety and efficacy of the slow rate release paclitaxel-eluting TAXUS™ stent compared to an otherwise identical uncoated bare metal EXPRESS2™ stent.

DETAILED DESCRIPTION:
Prospective, 2 x 2 factorial single blind, randomized, multi-center trial of 3400 patients enrolled at up to 200 centers. Patients will be randomized 1:1 in the emergency room to a) anticoagulation with unfractionated heparin plus routine GP IIb/IIIa inhibition vs. b) bivalirudin and bail-out GP IIb/IIIa inhibition. Following angiography, patients with lesions eligible for stenting will then undergo a second randomization (3:1) to stent implantation with either a) a slow rate-release paclitaxel-eluting stent (TAXUS™) or b) an otherwise identical uncoated bare metal stent (EXPRESS2™).

ELIGIBILITY:
Inclusion Criteria:

* Must have clinical symptoms consistent with AMI (e.g., angina or anginal equivalent)lasting >20 minutes but <12 hours in duration;
* ST-segment elevation of >1 mm in >2 contiguous leads, or (presumably new) left bundle branch block, or true posterior MI with ST depression of >1 mm in >2 contiguous anterior leads;
* The patient or guardian agrees to the study protocol and the schedule of clinical and angiographic follow-up, and provides informed, written consent.

Exclusion Criteria:

* The patient has a known hypersensitivity or contraindication to any of the following medications:

  * Heparin, pork or pork products
  * Both abciximab and eptifibatide
  * Aspirin
  * Both Clopidogrel and Ticlopidine
  * Bivalirudin
  * Paclitaxel or Taxol
  * The polymer components of the TAXUS™ stent (SIBS)
  * Stainless steel and/or
  * Contrast media;
* Prior administration of thrombolytic therapy, bivalirudin, GP IIb/IIIa inhibitors, low molecular weight heparin or fondaparinux for this admission. Patients receiving prior unfractionated heparin may be enrolled, and treated per randomization;
* Current use of coumadin;
* Systemic (intravenous) Paclitaxel or Taxol use within 12 months;
* Female of childbearing potential, unless a recent pregnancy test is negative, who possibly plans to become pregnant any time after enrollment into this study;
* History of bleeding diathesis or known coagulopathy (including heparin-induced thrombocytopenia), or will refuse blood transfusions;
* History of intra-cerebral mass, aneurysm, arteriovenous malformation, or hemorrhagic stroke;
* Stroke or transient ischemic attack within the past 6 months, or any permanent residual neurologic defect;
* Gastrointestinal or genitourinary bleeding within the last 2 months, or major surgery within six weeks;
* Recent history or known current platelet count <100,000 cells/mm3 or Hgb <10 g/dL;
* Extensive peripheral vascular disease, such that emergent angiography and intervention in the opinion of the investigator is likely to be difficult or complicated;
* An elective surgical procedure is planned that would necessitate interruption of thienopyridines during the first six months post enrollment;
* Non-cardiac co-morbid conditions are present with life expectancy <1 year or that may result in protocol non-compliance;
* Patients who are actively participating in another drug or device investigational study, which have not completed the primary endpoint follow-up period;
* Previous enrollment in this trial;
* Patients who underwent coronary stent implantation within the past 30 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3602 (Actual)
Dates: Start 2005-03; Primary Completion 2008-06 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregg W Stone, MD, Principal Investigator — CardioVascular Research Foundation; Roxana Mehran, MD, Study Director — CardioVascular Research Foundation
Locations (1):
- LeBauer CV Research Foundation, Greensboro, North Carolina, United States

REFERENCES:
- [Derived] Kosmidou I, McAndrew T, Redfors B, Embacher M, Dizon JM, Mehran R, Ben-Yehuda O, Mintz GS, Stone GW. Correlation of Admission Heart Rate With Angiographic and Clinical Outcomes in Patients With Right Coronary Artery ST-Segment Elevation Myocardial Infarction Undergoing Primary Percutaneous Coronary Intervention: HORIZONS-AMI (The Harmonizing Outcomes With Revascularization and Stents in Acute Myocardial Infarction) Trial. J Am Heart Assoc. 2017 Jul 19;6(7):e006181. doi: 10.1161/JAHA.117.006181. PMID 28724652
- [Derived] Tamez H, Pinto DS, Kirtane AJ, Litherland C, Yeh RW, Dangas GD, Mehran R, Deliargyris EN, Ortiz G, Gibson CM, Stone GW. Effect of Short Procedural Duration With Bivalirudin on Increased Risk of Acute Stent Thrombosis in Patients With STEMI: A Secondary Analysis of the HORIZONS-AMI Randomized Clinical Trial. JAMA Cardiol. 2017 Jun 1;2(6):673-677. doi: 10.1001/jamacardio.2016.5669. PMID 28249084
- [Derived] Ducrocq G, Steg PG, Van't Hof A, Zeymer U, Mehran R, Hamm CW, Bernstein D, Prats J, Deliargyris EN, Stone GW. Utility of post-procedural anticoagulation after primary PCI for STEMI: insights from a pooled analysis of the HORIZONS-AMI and EUROMAX trials. Eur Heart J Acute Cardiovasc Care. 2017 Oct;6(7):659-665. doi: 10.1177/2048872616650869. Epub 2016 Jun 10. PMID 27287251
- [Derived] Dangas GD, Schoos MM, Steg PG, Mehran R, Clemmensen P, van 't Hof A, Prats J, Bernstein D, Deliargyris EN, Stone GW. Early Stent Thrombosis and Mortality After Primary Percutaneous Coronary Intervention in ST-Segment-Elevation Myocardial Infarction: A Patient-Level Analysis of 2 Randomized Trials. Circ Cardiovasc Interv. 2016 May;9(5):e003272. doi: 10.1161/CIRCINTERVENTIONS.115.003272. PMID 27165710
- [Derived] Weisz G, Smilowitz NR, Kirtane AJ, Rinaldi MJ, Parvataneni R, Xu K, Stuckey TD, Maehara A, Witzenbichler B, Neumann FJ, Metzger DC, Henry TD, Cox DA, Duffy PL, Brodie BR, Mazzaferri EL Jr, Mehran R, Stone GW. Proton Pump Inhibitors, Platelet Reactivity, and Cardiovascular Outcomes After Drug-Eluting Stents in Clopidogrel-Treated Patients: The ADAPT-DES Study. Circ Cardiovasc Interv. 2015 Oct;8(10):e001952. doi: 10.1161/CIRCINTERVENTIONS.114.001952. PMID 26458411
- [Derived] Giacoppo D, Madhavan MV, Baber U, Warren J, Bansilal S, Witzenbichler B, Dangas GD, Kirtane AJ, Xu K, Kornowski R, Brener SJ, Genereux P, Stone GW, Mehran R. Impact of Contrast-Induced Acute Kidney Injury After Percutaneous Coronary Intervention on Short- and Long-Term Outcomes: Pooled Analysis From the HORIZONS-AMI and ACUITY Trials. Circ Cardiovasc Interv. 2015 Aug;8(8):e002475. doi: 10.1161/CIRCINTERVENTIONS.114.002475. PMID 26198286
- [Derived] Nikolsky E, Mehran R, Dangas GD, Xu K, Parvataneni R, Witzenbichler B, Guagliumi G, Kornowski R, Genereux P, Brener SJ, Stone GW. Cerebrovascular events after a primary percutaneous coronary intervention strategy for acute ST-segment-elevation myocardial infarction: analysis from the HORIZONS-AMI Trial. Circ Cardiovasc Interv. 2015 Apr;8(4):e002283. doi: 10.1161/CIRCINTERVENTIONS.114.002283. PMID 25858976
- [Derived] Stone GW, Mehran R, Goldstein P, Witzenbichler B, Van't Hof A, Guagliumi G, Hamm CW, Genereux P, Clemmensen P, Pocock SJ, Gersh BJ, Bernstein D, Deliargyris EN, Steg PG. Bivalirudin versus heparin with or without glycoprotein IIb/IIIa inhibitors in patients with STEMI undergoing primary percutaneous coronary intervention: pooled patient-level analysis from the HORIZONS-AMI and EUROMAX trials. J Am Coll Cardiol. 2015 Jan 6;65(1):27-38. doi: 10.1016/j.jacc.2014.10.029. PMID 25572507
- [Derived] Sanborn TA, Tomey MI, Mehran R, Genereux P, Witzenbichler B, Brener SJ, Kirtane AJ, McAndrew TC, Kornowski R, Dudek D, Nikolsky E, Stone GW. Femoral vascular closure device use, bivalirudin anticoagulation, and bleeding after primary angioplasty for STEMI: results from the HORIZONS-AMI trial. Catheter Cardiovasc Interv. 2015 Feb 15;85(3):371-9. doi: 10.1002/ccd.25663. Epub 2014 Oct 28. PMID 25179260
- [Derived] Stone SG, Serrao GW, Mehran R, Tomey MI, Witzenbichler B, Guagliumi G, Peruga JZ, Brodie BR, Dudek D, Mockel M, Brener SJ, Dangas G, Stone GW. Incidence, predictors, and implications of reinfarction after primary percutaneous coronary intervention in ST-segment-elevation myocardial infarction: the Harmonizing Outcomes with Revascularization and Stents in Acute Myocardial Infarction Trial. Circ Cardiovasc Interv. 2014 Aug;7(4):543-51. doi: 10.1161/CIRCINTERVENTIONS.114.001360. Epub 2014 Jun 17. PMID 24939928
- [Derived] Keeley EC, Mehran R, Brener SJ, Witzenbichler B, Guagliumi G, Dudek D, Kornowski R, Dressler O, Fahy M, Xu K, Grines CL, Stone GW. Impact of multiple complex plaques on short- and long-term clinical outcomes in patients presenting with ST-segment elevation myocardial infarction (from the Harmonizing Outcomes With Revascularization and Stents in Acute Myocardial Infarction [HORIZONS-AMI] Trial). Am J Cardiol. 2014 May 15;113(10):1621-7. doi: 10.1016/j.amjcard.2014.02.016. Epub 2014 Mar 1. PMID 24703369
- [Derived] Larsen AI, Tomey MI, Mehran R, Nilsen DW, Kirtane AJ, Witzenbichler B, Guagliumi G, Brener SJ, Genereux P, Kornowski R, Dudek D, Gersh BJ, Stone GW. Comparison of outcomes in patients with ST-segment elevation myocardial infarction discharged on versus not on statin therapy (from the Harmonizing Outcomes With Revascularization and Stents in Acute Myocardial Infarction Trial). Am J Cardiol. 2014 Apr 15;113(8):1273-9. doi: 10.1016/j.amjcard.2014.01.401. Epub 2014 Jan 31. PMID 24576541
- [Derived] Genereux P, Madhavan MV, Mintz GS, Maehara A, Palmerini T, Lasalle L, Xu K, McAndrew T, Kirtane A, Lansky AJ, Brener SJ, Mehran R, Stone GW. Ischemic outcomes after coronary intervention of calcified vessels in acute coronary syndromes. Pooled analysis from the HORIZONS-AMI (Harmonizing Outcomes With Revascularization and Stents in Acute Myocardial Infarction) and ACUITY (Acute Catheterization and Urgent Intervention Triage Strategy) TRIALS. J Am Coll Cardiol. 2014 May 13;63(18):1845-54. doi: 10.1016/j.jacc.2014.01.034. Epub 2014 Feb 19. PMID 24561145
- [Derived] Stone GW, Clayton T, Deliargyris EN, Prats J, Mehran R, Pocock SJ. Reduction in cardiac mortality with bivalirudin in patients with and without major bleeding: The HORIZONS-AMI trial (Harmonizing Outcomes with Revascularization and Stents in Acute Myocardial Infarction). J Am Coll Cardiol. 2014 Jan 7-14;63(1):15-20. doi: 10.1016/j.jacc.2013.09.027. Epub 2013 Oct 16. PMID 24140664
- [Derived] Brener SJ, Dizon JM, Mehran R, Guerchicoff A, Lansky AJ, Farkouh M, Brodie B, Guagliumi G, Witzenbichler B, Fahy M, Parise H, Stone GW. Complementary prognostic utility of myocardial blush grade and ST-segment resolution after primary percutaneous coronary intervention: analysis from the HORIZONS-AMI trial. Am Heart J. 2013 Oct;166(4):676-83. doi: 10.1016/j.ahj.2013.07.025. Epub 2013 Sep 13. PMID 24093847
- [Derived] Palmerini T, Brener SJ, Mehran R, Dangas G, Genereux P, Riva DD, Mariani A, Xu K, Stone GW. Leukocyte count is a modulating factor for the mortality benefit of bivalirudin in ST-segment-elevation acute myocardial infarction: the HORIZONS-AMI trial. Circ Cardiovasc Interv. 2013 Oct 1;6(5):518-26. doi: 10.1161/CIRCINTERVENTIONS.113.000592. Epub 2013 Oct 1. PMID 24084625
- [Derived] Farkouh ME, Reiffel J, Dressler O, Nikolsky E, Parise H, Cristea E, Baran DA, Dizon J, Merab JP, Lansky AJ, Mehran R, Stone GW. Relationship between ST-segment recovery and clinical outcomes after primary percutaneous coronary intervention: the HORIZONS-AMI ECG substudy report. Circ Cardiovasc Interv. 2013 Jun;6(3):216-23. doi: 10.1161/CIRCINTERVENTIONS.112.000142. Epub 2013 May 7. PMID 23652600
- [Derived] Rakowski T, Dudek D, Dziewierz A, Yu J, Witzenbichler B, Guagliumi G, Kornowski R, Hartmann F, Lansky AJ, Brener SJ, Mehran R, Stone GW. Impact of infarct-related artery patency before primary PCI on outcome in patients with ST-segment elevation myocardial infarction: the HORIZONS-AMI trial. EuroIntervention. 2013 Mar;8(11):1307-14. doi: 10.4244/EIJV8I11A199. PMID 23538158
- [Derived] Caixeta A, Lansky AJ, Mehran R, Brener SJ, Claessen B, Genereux P, Palmerini T, Witzenbichler B, Guagliumi G, Brodie BR, Dudek D, Fahy M, Dangas GD, Stone GW; Harmonizing Outcomes With Revascularization and Stents in Acute Myocardial Infarction (HORIZONS-AMI) trial investigators. Predictors of suboptimal TIMI flow after primary angioplasty for acute myocardial infarction: results from the HORIZONS-AMI trial. EuroIntervention. 2013 Jun 22;9(2):220-7. doi: 10.4244/EIJV9I2A37. PMID 23518872
- [Derived] Tobbia P, Brodie BR, Witzenbichler B, Metzger C, Guagliumi G, Yu J, Kellett MA, Stuckey T, Fahy M, Mehran R, Stone GW. Adverse event rates following primary PCI for STEMI at US and non-US hospitals: three-year analysis from the HORIZONS-AMI trial. EuroIntervention. 2013 Feb 22;8(10):1134-42. doi: 10.4244/EIJV8I10A176. PMID 23425539
- [Derived] Dudek D, Mehran R, Dziewierz A, Witzenbichler B, Brodie BR, Kornowski R, Fahy M, Lansky AJ, Rakowski T, Legutko J, Bryniarski L, Stone GW. Impact of advanced age on the safety and effectiveness of paclitaxel-eluting stent implantation in patients with ST-segment elevation myocardial infarction undergoing primary angioplasty: The HORIZONS-AMI trial. Catheter Cardiovasc Interv. 2013 Nov 15;82(6):869-77. doi: 10.1002/ccd.24813. Epub 2013 Aug 1. PMID 23359554
- [Derived] Dangas GD, Claessen BE, Mehran R, Xu K, Stone GW. Stent thrombosis after primary angioplasty for STEMI in relation to non-adherence to dual antiplatelet therapy over time: results of the HORIZONS-AMI trial. EuroIntervention. 2013 Jan 22;8(9):1033-9. doi: 10.4244/EIJV8I9A159. PMID 23339809
- [Derived] Zhao Z, Witzenbichler B, Mintz GS, Jaster M, Choi SY, Wu X, He Y, Margolis MP, Dressler O, Cristea E, Parise H, Mehran R, Stone GW, Maehara A. Dynamic nature of nonculprit coronary artery lesion morphology in STEMI: a serial IVUS analysis from the HORIZONS-AMI trial. JACC Cardiovasc Imaging. 2013 Jan;6(1):86-95. doi: 10.1016/j.jcmg.2012.08.010. PMID 23328566
- [Derived] Jarai R, Dangas G, Huber K, Xu K, Brodie BR, Witzenbichler B, Metzger DC, Radke PW, Yu J, Claessen BE, Genereux P, Mehran R, Stone GW. B-type natriuretic peptide and risk of contrast-induced acute kidney injury in acute ST-segment-elevation myocardial infarction: a substudy from the HORIZONS-AMI trial. Circ Cardiovasc Interv. 2012 Dec;5(6):813-20. doi: 10.1161/CIRCINTERVENTIONS.112.972356. Epub 2012 Nov 27. PMID 23192919
- [Derived] Dangas GD, Claessen BE, Mehran R, Xu K, Fahy M, Parise H, Henriques JP, Ohman EM, White HD, Stone GW. Development and validation of a stent thrombosis risk score in patients with acute coronary syndromes. JACC Cardiovasc Interv. 2012 Nov;5(11):1097-105. doi: 10.1016/j.jcin.2012.07.012. PMID 23174632
- [Derived] Planer D, Witzenbichler B, Guagliumi G, Peruga JZ, Brodie BR, Xu K, Fahy M, Mehran R, Stone GW. Impact of hyperglycemia in patients with ST-segment elevation myocardial infarction undergoing percutaneous coronary intervention: the HORIZONS-AMI trial. Int J Cardiol. 2013 Sep 10;167(6):2572-9. doi: 10.1016/j.ijcard.2012.06.054. Epub 2012 Jul 12. PMID 22795245
- [Derived] Dangas GD, Claessen BE, Mehran R, Brener S, Brodie BR, Dudek D, Witzenbichler B, Peruga JZ, Guagliumi G, Moses JW, Lansky AJ, Xu K, Stone GW. Clinical outcomes following stent thrombosis occurring in-hospital versus out-of-hospital: results from the HORIZONS-AMI (Harmonizing Outcomes with Revascularization and Stents in Acute Myocardial Infarction) trial. J Am Coll Cardiol. 2012 May 15;59(20):1752-9. doi: 10.1016/j.jacc.2011.12.042. PMID 22575312
- [Derived] Xu K, Mintz GS, Kubo T, Wu X, Guo N, Yang J, Witzenbichler B, Guagliumi G, Brodie B, Dressler O, Cristea E, Parise H, Mehran R, Stone GW, Maehara A. Long-term follow-up of attenuated plaques in patients with acute myocardial infarction: an intravascular ultrasound substudy of the HORIZONS-AMI trial. Circ Cardiovasc Interv. 2012 Apr;5(2):185-92. doi: 10.1161/CIRCINTERVENTIONS.111.964684. Epub 2012 Mar 20. PMID 22438429
- [Derived] Suh JW, Mehran R, Claessen BE, Xu K, Baber U, Dangas G, Parise H, Lansky AJ, Witzenbichler B, Grines CL, Guagliumi G, Kornowski R, Wohrle J, Dudek D, Weisz G, Stone GW. Impact of in-hospital major bleeding on late clinical outcomes after primary percutaneous coronary intervention in acute myocardial infarction the HORIZONS-AMI (Harmonizing Outcomes With Revascularization and Stents in Acute Myocardial Infarction) trial. J Am Coll Cardiol. 2011 Oct 18;58(17):1750-6. doi: 10.1016/j.jacc.2011.07.021. PMID 21996385
- [Derived] Kornowski R, Mehran R, Dangas G, Nikolsky E, Assali A, Claessen BE, Gersh BJ, Wong SC, Witzenbichler B, Guagliumi G, Dudek D, Fahy M, Lansky AJ, Stone GW; HORIZONS-AMI Trial Investigators. Prognostic impact of staged versus "one-time" multivessel percutaneous intervention in acute myocardial infarction: analysis from the HORIZONS-AMI (harmonizing outcomes with revascularization and stents in acute myocardial infarction) trial. J Am Coll Cardiol. 2011 Aug 9;58(7):704-11. doi: 10.1016/j.jacc.2011.02.071. PMID 21816305
- [Derived] Witzenbichler B, Mehran R, Guagliumi G, Dudek D, Huber K, Kornowski R, Stuckey TD, Fahy M, Parise H, Stone GW. Impact of diabetes mellitus on the safety and effectiveness of bivalirudin in patients with acute myocardial infarction undergoing primary angioplasty: analysis from the HORIZONS-AMI (Harmonizing Outcomes with RevasculariZatiON and Stents in Acute Myocardial Infarction) trial. JACC Cardiovasc Interv. 2011 Jul;4(7):760-8. doi: 10.1016/j.jcin.2011.04.008. PMID 21777884
- [Derived] Stone GW, Witzenbichler B, Guagliumi G, Peruga JZ, Brodie BR, Dudek D, Kornowski R, Hartmann F, Gersh BJ, Pocock SJ, Dangas G, Wong SC, Fahy M, Parise H, Mehran R; HORIZONS-AMI Trial Investigators. Heparin plus a glycoprotein IIb/IIIa inhibitor versus bivalirudin monotherapy and paclitaxel-eluting stents versus bare-metal stents in acute myocardial infarction (HORIZONS-AMI): final 3-year results from a multicentre, randomised controlled trial. Lancet. 2011 Jun 25;377(9784):2193-204. doi: 10.1016/S0140-6736(11)60764-2. Epub 2011 Jun 12. PMID 21665265
- [Derived] Palmerini T, Mehran R, Dangas G, Nikolsky E, Witzenbichler B, Guagliumi G, Dudek D, Genereux P, Caixeta A, Rabbani L, Weisz G, Parise H, Fahy M, Xu K, Brodie B, Lansky A, Stone GW. Impact of leukocyte count on mortality and bleeding in patients with myocardial infarction undergoing primary percutaneous coronary interventions: analysis from the Harmonizing Outcome with Revascularization and Stent in Acute Myocardial Infarction trial. Circulation. 2011 Jun 21;123(24):2829-37, 7 p following 2837. doi: 10.1161/CIRCULATIONAHA.110.985564. Epub 2011 May 31. PMID 21632496
- [Derived] Wu X, Mintz GS, Xu K, Lansky AJ, Witzenbichler B, Guagliumi G, Brodie B, Kellett MA Jr, Dressler O, Parise H, Mehran R, Stone GW, Maehara A. The relationship between attenuated plaque identified by intravascular ultrasound and no-reflow after stenting in acute myocardial infarction: the HORIZONS-AMI (Harmonizing Outcomes With Revascularization and Stents in Acute Myocardial Infarction) trial. JACC Cardiovasc Interv. 2011 May;4(5):495-502. doi: 10.1016/j.jcin.2010.12.012. PMID 21596321
- [Derived] Choi SY, Witzenbichler B, Maehara A, Lansky AJ, Guagliumi G, Brodie B, Kellett MA Jr, Dressler O, Parise H, Mehran R, Dangas GD, Mintz GS, Stone GW. Intravascular ultrasound findings of early stent thrombosis after primary percutaneous intervention in acute myocardial infarction: a Harmonizing Outcomes with Revascularization and Stents in Acute Myocardial Infarction (HORIZONS-AMI) substudy. Circ Cardiovasc Interv. 2011 Jun;4(3):239-47. doi: 10.1161/CIRCINTERVENTIONS.110.959791. Epub 2011 May 17. PMID 21586693
- [Derived] Dangas GD, Caixeta A, Mehran R, Parise H, Lansky AJ, Cristea E, Brodie BR, Witzenbichler B, Guagliumi G, Peruga JZ, Dudek D, Moeckel M, Stone GW; Harmonizing Outcomes With Revascularization and Stents in Acute Myocardial Infarction (HORIZONS-AMI) Trial Investigators. Frequency and predictors of stent thrombosis after percutaneous coronary intervention in acute myocardial infarction. Circulation. 2011 Apr 26;123(16):1745-56. doi: 10.1161/CIRCULATIONAHA.110.981688. Epub 2011 Apr 11. PMID 21482968
- [Derived] Witzenbichler B, Wohrle J, Guagliumi G, Peruga JZ, Brodie BR, Dudek D, Kornowski R, Hartmann F, Hood KL, Parise H, Lansky AJ, Nikolsky E, Mehran R, Stone GW. Paclitaxel-eluting stents compared with bare metal stents in diabetic patients with acute myocardial infarction: the Harmonizing Outcomes with Revascularization and Stents in Acute Myocardial Infarction (HORIZONS-AMI) trial. Circ Cardiovasc Interv. 2011 Apr 1;4(2):130-8. doi: 10.1161/CIRCINTERVENTIONS.110.960245. Epub 2011 Mar 1. PMID 21364152
- [Derived] Hakim DA, Dangas GD, Caixeta A, Nikolsky E, Lansky AJ, Moses JW, Claessen B, Sanidas E, White HD, Ohman EM, Manoukian SV, Fahy M, Mehran R, Stone GW. Impact of baseline thrombocytopenia on the early and late outcomes after ST-elevation myocardial infarction treated with primary angioplasty: analysis from the Harmonizing Outcomes with Revascularization and Stents in Acute Myocardial Infarction (HORIZONS-AMI) trial. Am Heart J. 2011 Feb;161(2):391-6. doi: 10.1016/j.ahj.2010.11.001. PMID 21315224
- [Derived] Guagliumi G, Costa MA, Sirbu V, Musumeci G, Bezerra HG, Suzuki N, Matiashvili A, Lortkipanidze N, Mihalcsik L, Trivisonno A, Valsecchi O, Mintz GS, Dressler O, Parise H, Maehara A, Cristea E, Lansky AJ, Mehran R, Stone GW. Strut coverage and late malapposition with paclitaxel-eluting stents compared with bare metal stents in acute myocardial infarction: optical coherence tomography substudy of the Harmonizing Outcomes with Revascularization and Stents in Acute Myocardial Infarction (HORIZONS-AMI) Trial. Circulation. 2011 Jan 25;123(3):274-81. doi: 10.1161/CIRCULATIONAHA.110.963181. Epub 2011 Jan 10. PMID 21220730
- [Derived] Stone GW, Parise H, Witzenbichler B, Kirtane A, Guagliumi G, Peruga JZ, Brodie BR, Dudek D, Mockel M, Lansky AJ, Mehran R. Selection criteria for drug-eluting versus bare-metal stents and the impact of routine angiographic follow-up: 2-year insights from the HORIZONS-AMI (Harmonizing Outcomes With Revascularization and Stents in Acute Myocardial Infarction) trial. J Am Coll Cardiol. 2010 Nov 2;56(19):1597-604. doi: 10.1016/j.jacc.2010.08.608. Epub 2010 Oct 1. PMID 20888162
- [Derived] Guo N, Maehara A, Mintz GS, He Y, Xu K, Wu X, Lansky AJ, Witzenbichler B, Guagliumi G, Brodie B, Kellett MA Jr, Dressler O, Parise H, Mehran R, Stone GW. Incidence, mechanisms, predictors, and clinical impact of acute and late stent malapposition after primary intervention in patients with acute myocardial infarction: an intravascular ultrasound substudy of the Harmonizing Outcomes with Revascularization and Stents in Acute Myocardial Infarction (HORIZONS-AMI) trial. Circulation. 2010 Sep 14;122(11):1077-84. doi: 10.1161/CIRCULATIONAHA.109.906040. Epub 2010 Aug 30. PMID 20805433
- [Derived] Parodi G, Antoniucci D, Nikolsky E, Witzenbichler B, Guagliumi G, Peruga JZ, Stuckey T, Dudek D, Kornowski R, Hartmann F, Lansky AJ, Mehran R, Stone GW. Impact of bivalirudin therapy in high-risk patients with acute myocardial infarction: 1-year results from the HORIZONS-AMI (Harmonizing Outcomes with RevasculariZatiON and Stents in Acute Myocardial Infarction) trial. JACC Cardiovasc Interv. 2010 Aug;3(8):796-802. doi: 10.1016/j.jcin.2010.05.009. PMID 20723849
- [Derived] Maehara A, Mintz GS, Lansky AJ, Witzenbichler B, Guagliumi G, Brodie B, Kellett MA Jr, Parise H, Mehran R, Stone GW. Volumetric intravascular ultrasound analysis of Paclitaxel-eluting and bare metal stents in acute myocardial infarction: the harmonizing outcomes with revascularization and stents in acute myocardial infarction intravascular ultrasound substudy. Circulation. 2009 Nov 10;120(19):1875-82. doi: 10.1161/CIRCULATIONAHA.109.873893. Epub 2009 Oct 26. PMID 19858413
- [Derived] Dangas G, Mehran R, Guagliumi G, Caixeta A, Witzenbichler B, Aoki J, Peruga JZ, Brodie BR, Dudek D, Kornowski R, Rabbani LE, Parise H, Stone GW; HORIZONS-AMI Trial Investigators. Role of clopidogrel loading dose in patients with ST-segment elevation myocardial infarction undergoing primary angioplasty: results from the HORIZONS-AMI (harmonizing outcomes with revascularization and stents in acute myocardial infarction) trial. J Am Coll Cardiol. 2009 Oct 6;54(15):1438-46. doi: 10.1016/j.jacc.2009.06.021. PMID 19796737
- [Derived] Mehran R, Lansky AJ, Witzenbichler B, Guagliumi G, Peruga JZ, Brodie BR, Dudek D, Kornowski R, Hartmann F, Gersh BJ, Pocock SJ, Wong SC, Nikolsky E, Gambone L, Vandertie L, Parise H, Dangas GD, Stone GW; HORIZONS-AMI Trial Investigators. Bivalirudin in patients undergoing primary angioplasty for acute myocardial infarction (HORIZONS-AMI): 1-year results of a randomised controlled trial. Lancet. 2009 Oct 3;374(9696):1149-59. doi: 10.1016/S0140-6736(09)61484-7. Epub 2009 Aug 28. PMID 19717185
- [Derived] Stone GW, Lansky AJ, Pocock SJ, Gersh BJ, Dangas G, Wong SC, Witzenbichler B, Guagliumi G, Peruga JZ, Brodie BR, Dudek D, Mockel M, Ochala A, Kellock A, Parise H, Mehran R; HORIZONS-AMI Trial Investigators. Paclitaxel-eluting stents versus bare-metal stents in acute myocardial infarction. N Engl J Med. 2009 May 7;360(19):1946-59. doi: 10.1056/NEJMoa0810116. PMID 19420364
- [Derived] Mehran R, Brodie B, Cox DA, Grines CL, Rutherford B, Bhatt DL, Dangas G, Feit F, Ohman EM, Parise H, Fahy M, Lansky AJ, Stone GW. The Harmonizing Outcomes with RevasculariZatiON and Stents in Acute Myocardial Infarction (HORIZONS-AMI) Trial: study design and rationale. Am Heart J. 2008 Jul;156(1):44-56. doi: 10.1016/j.ahj.2008.02.008. PMID 18585496
- [Derived] Stone GW, Witzenbichler B, Guagliumi G, Peruga JZ, Brodie BR, Dudek D, Kornowski R, Hartmann F, Gersh BJ, Pocock SJ, Dangas G, Wong SC, Kirtane AJ, Parise H, Mehran R; HORIZONS-AMI Trial Investigators. Bivalirudin during primary PCI in acute myocardial infarction. N Engl J Med. 2008 May 22;358(21):2218-30. doi: 10.1056/NEJMoa0708191. PMID 18499566

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between March 25, 2005, and May 7, 2007, 3602 patients with STEMI undergoing primary percutaneous coronary intervention were enrolled at 123 academic or community-based medical centers in 11 countries.
Pre-assignment Details: Random, open-label assignment (1:1 ratio) to unfractionated heparin plus a glycoprotein IIb/IIIa inhibitor or bivalirudin alone. After emergency angiography and triage to PCI, CABG, or GDMT, eligible patients were randomly assigned (3:1 ratio) to either paclitaxel-eluting stents or uncoated, bare-metal stents.
Groups:
- Pharmacology Arm - Bivalirudin; Pharmacology Arm - Unfractionated Heparin: To establish the safety and efficacy of the use of bivalirudin in patients with acute myocardial infarction undergoing a primary angioplasty strategy by showing that compared to unfractionated heparin plus routine use of GP IIb/IIIa inhibitors, bivalirudin (with use of GP IIb/IIIa inhibitors reserved for angioplasty complications) results in:
  1. reduced rates of major bleeding events at 30 days
  2. similar rates of major adverse ischemic cardiac events at 30 days
  3. reduced rates of the composite of major adverse ischemic cardiac events + major bleeding at 30 days.
  Bivalirudin: Bivalirudin bolus of 0.75 mg/kg IV, followed by an infusion of 1.75 mg/kg/h as soon as logistically feasible (ideally in the emergency room).
  Unfractionated heparin: 60 U/kg of IV heparin, started as soon as possible (ideally in the emergency room).
- Stent Arm - Paclitaxel-Eluting Stent; Stent Arm - Bare Metal Stent: To establish the safety and efficacy of the paclitaxel-eluting TAXUS™ stent by showing that compared to an otherwise identical bare metal EXPRESS2™ stent, the TAXUS™ stent results in:
  1. reduced rates of target lesion revascularization for ischemia at 1 year
  2. similar rates of death, reinfarction, stroke or stent thrombosis at 1 year
  3. lower rates of analysis segment binary angiographic restenosis at 13 months
  Bare metal stent: Uncoated bare metal stent
  Paclitaxel-eluting stent: slow rate-release paclitaxel-eluting stent
Period: Pharmacology Intervention/Randomization
Arm/Group | Pharmacology Arm - Bivalirudin | Pharmacology Arm - Unfractionated Heparin | Stent Arm - Paclitaxel-Eluting Stent | Stent Arm - Bare Metal Stent
Started | 1800 | 1802 | 0 | 0
30-Day Follow-up | 1787 | 1791 | 0 | 0
1-Year Follow-up | 1696 | 1702 | 0 | 0
3-Year Follow-up | 1634 | 1628 | 0 | 0
Completed | 1634 | 1628 | 0 | 0
Not Completed | 166 | 174 | 0 | 0
Not completed — Withdrawal by Subject | 40 | 43 | 0 | 0
Not completed — Lost to Follow-up | 97 | 103 | 0 | 0
Not completed — Not true myocardial infarction | 29 | 28 | 0 | 0
Period: Stent Intervention/Randomization
Arm/Group | Pharmacology Arm - Bivalirudin | Pharmacology Arm - Unfractionated Heparin | Stent Arm - Paclitaxel-Eluting Stent | Stent Arm - Bare Metal Stent
Started | 0 | 0 | 2257 | 749
1-Year Follow-up | 0 | 0 | 2186 | 715
3-Year Follow-up | 0 | 0 | 2103 | 687
Completed | 0 | 0 | 2103 | 687
Not Completed | 0 | 0 | 154 | 62
Not completed — Withdrawal by Subject | 0 | 0 | 41 | 15
Not completed — Lost to Follow-up | 0 | 0 | 113 | 47

BASELINE CHARACTERISTICS:
Population: Baseline data is presented by first randomization (pharmacology).
Groups:
- Total: Total of all reporting groups
Arm/Group | Pharmacology Arm - Bivalirudin | Pharmacology Arm - Unfractionated Heparin | Total
Number analyzed (Participants) | 1800 | 1802 | 3602
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 59.8 [51.9 to 69.5] | 60.7 [52.9 to 70.1] | 60.2 [52.4 to 69.9]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 412 | 430 | 842
  Male | 1388 | 1372 | 2760

OUTCOME MEASURES:

1. Primary Outcome: Pharmacology Arm - Major Adverse Ischemic Cardiac Events and Major Bleeding Events
Description: Number of participants with major adverse cardiovascular events (death, reinfarction, target-vessel revascularization for ischemia, and stroke) and major bleeding (bleeding adjudicated as not related to coronary artery bypass grafting).
Time Frame: 30 Days
Measure: Count of Participants; unit: Participants
Arm/Group | Pharmacology Arm - Bivalirudin | Pharmacology Arm - Unfractionated Heparin
Number analyzed (Participants) | 1800 | 1802
Participants | 166 | 218

2. Primary Outcome: Stent Arm - Ischemic Target Lesion Revascularization
Description: Number of Participants With Ischemic Target Lesion Revascularization
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Stent Arm - Paclitaxel-Eluting Stent | Stent Arm - Bare Metal Stent
Number analyzed (Participants) | 2257 | 749
Participants | 98 | 54

3. Primary Outcome: Stent Arm - Death, Reinfarction, Stroke, or Stent Thrombosis
Description: Number of Participants With Death, Reinfarction, Stroke, or Stent Thrombosis
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Stent Arm - Paclitaxel-Eluting Stent | Stent Arm - Bare Metal Stent
Number analyzed (Participants) | 2257 | 749
Participants | 181 | 59

4. Secondary Outcome: Pharmacology Arm - Major Adverse Cardiovascular Events
Description: Number of participants with major adverse cardiovascular events (death, reinfarction, target-vessel revascularization for ischemia, and stroke)
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Pharmacology Arm - Bivalirudin | Pharmacology Arm - Unfractionated Heparin
Number analyzed (Participants) | 1800 | 1802
Participants | 98 | 99

5. Secondary Outcome: Pharmacology Arm - Non-Coronary Artery Bypass Grafting-Related Major Bleeding
Description: Number of participants with major bleeding (bleeding adjudicated as not related to coronary artery bypass grafting)
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Pharmacology Arm - Bivalirudin | Pharmacology Arm - Unfractionated Heparin
Number analyzed (Participants) | 1800 | 1802
Participants | 89 | 149

6. Secondary Outcome: Stent Arm - Segment Binary Angiographic Restenosis
Description: Number of Participants With Segment Binary Angiographic Restenosis (13-month Angiographic Subset).
Time Frame: 13 months
Measure: Count of Participants; unit: Participants
Arm/Group | Stent Arm - Paclitaxel-Eluting Stent | Stent Arm - Bare Metal Stent
Number analyzed (Participants) | 1062 | 328
Participants | 102 | 76

7. Secondary Outcome: Pharmacology Arm - Major Adverse Cardiovascular Events
Description: as for outcome 4
Time Frame: 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | Pharmacology Arm - Bivalirudin | Pharmacology Arm - Unfractionated Heparin
Number analyzed (Participants) | 1800 | 1802
Participants | 379 | 377

ADVERSE EVENTS:
Time Frame: 3 Years
Arm/Group | Pharmacology Arm - Bivalirudin | Pharmacology Arm - Unfractionated Heparin | Stent Arm - Paclitaxel-Eluting Stent | Stent Arm - Bare Metal Stent
All-Cause Mortality (participants affected / at risk) | 102/1800 | 134/1802 | 123/2257 | 48/749
Serious Adverse Events (participants affected / at risk) | 397/1800 | 439/1802 | 473/2257 | 185/749
Other Adverse Events (participants affected / at risk) | 81/1800 | 132/1802 | 122/2257 | 32/749
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pharmacology Arm - Bivalirudin (N=1800) | Pharmacology Arm - Unfractionated Heparin (N=1802) | Stent Arm - Paclitaxel-Eluting Stent (N=2257) | Stent Arm - Bare Metal Stent (N=749)
Death (cardiac) (Cardiac disorders) | 50 (50) | 88 (88) | 71 (71) | 28 (28)
Stent thrombosis (definite or probable) (Cardiac disorders) | 75 (83) | 81 (88) | 110 (121) | 32 (34) — According to the Academic Research Consortium classification
Ischemia-driven target vessel revascularization (TVR) (Cardiac disorders) | 239 (272) | 200 (238) | 268 (303) | 126 (150)
Ischemia-driven target lesion revascularization (TLR) (Cardiac disorders) | 190 (215) | 160 (181) | 204 (228) | 108 (126)
Ischemia-driven TVR, non-TLR (Cardiac disorders) | 86 (94) | 68 (76) | 100 (105) | 38 (44)
Major bleeing (protocol), non-coronary artery bypass grafting-related (Cardiac disorders) | 121 (149) | 185 (207) | 189 (213) | 56 (68)
Blood transfusion (Cardiac disorders) | 91 (132) | 124 (150) | 105 (123) | 32 (43)
Thrombolysis in Myocardial Infarction (TIMI) major or minor bleeding (Cardiac disorders) | 124 (156) | 193 (212) | 165 (179) | 46 (55)
Global Use of Strategies to Open Occluded Arteries (GUSTO) Moderate Bleeding (Cardiac disorders) | 81 (120) | 110 (136) | 95 (112) | 29 (41)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pharmacology Arm - Bivalirudin (N=1800) | Pharmacology Arm - Unfractionated Heparin (N=1802) | Stent Arm - Paclitaxel-Eluting Stent (N=2257) | Stent Arm - Bare Metal Stent (N=749)
Thrombolysis in Myocardial Infarction Minor Bleeding (Cardiac disorders) | 57 (64) | 89 (91) | 85 (87) | 24 (26)
Global Use of Strategies to Open Occluded Arteries Mild Bleeding (Cardiac disorders) | 71 (71) | 110 (113) | 106 (109) | 28 (28)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No